CLINICAL TRIAL: NCT06569680
Title: Phase II Trial of Mosunetuzumab in Patients With Newly Diagnosed Extranodal Marginal Zone Lymphoma (EMZL) (ML44933)
Brief Title: Mosunetuzumab in Patients With Newly Diagnosed Extranodal Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Izidore Lossos, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Izidore Lossos, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240178
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Extranodal Marginal Zone Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mosunetuzumab Treatment Group (Experimental): Participants in this group will receive Mosunetuzumab for eight (8) 21-day cycles. Total participation is about 3.5 years.
  Interventions: Drug: Mosunetuzumab

INTERVENTIONS:
Drug: Mosunetuzumab — Mosunetuzumab will be administered via subcutaneous (SC) injection using a step-up dosing model. Participants will receive Mosunetuzumab on days 1, 8, and 15 of Cycle 1, and on day 1 of Cycles 2 through 8 as follows:
  * Cycle 1 Day 1: 5mg
  * Cycle 1 Day 8: 45mg
  * Cycle 1 Day 15: 45mg
  * Cycles 2 through 8, Day 1: 45mg
  Other Names: ML44933; Lunsumio; Mosunetuzumab-axgb

SUMMARY:
The purpose of this study is to test a new medication called Mosunetuzumab to see if it can help people with Extranodal Marginal Zone Lymphoma (EMZL). This study will include people who have not yet received any treatment for cancer and whose cancer is in stage I-IV. This study will help doctors understand if Mosunetuzumab improves outcomes in people with EMZL and if it is safe to use.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or older at the time of signing informed consent.
2. Able and willing to sign the informed consent form (ICF).
3. Ability to comply with the trial protocol.
4. Histologically confirmed EMZL presenting with stage I-IV disease.
5. Previously untreated participants.

   1. Participants with H. pylori-positive gastric EMZL who received an initial treatment with currently accepted antibiotics may be considered eligible if, after antibiotic regimen, participant has histologically confirmed MZL.
   2. Participants who were previously treated with localized therapy (eg, radiation or surgery) and never received systemic therapy and present with recurrent disease are eligible upon histological confirmation of MZL.
6. Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥1 lesion that measures >1.5 cm in the longest diameter (LDi) and ≥1.0 cm in the longest perpendicular diameter as assessed by CT or MRI, especially in extranodal sites, per response criteria for lymphomas (Cheson, et al., 2014). Imaging must be conducted within 6 weeks prior to the start of therapy.

   1. Participants with skin EMZL who do not meet the radiographically measurable disease criteria described herein are eligible for participation provided that skin lesion measures ≥1.5 cm in diameter by tape measure and is documented by photo or there are multiple skin lesions measuring >1 cm in diameter on the body and at least one of them is histologically confirmed as EMZL.
   2. Participants with gastric EMZL histologically confirmed and need therapy but do not have measurable disease and in which response to treatment can be assessed by multiple random gastric biopsies per Groupe d'Etude des Lymphomes de l'Adult (GELA) criteria (Ruskoné Fourmestraux, et al., 2011).
   3. Participants with conjunctival EMZL who do not meet the radiographically measurable disease criteria described herein are eligible for participation provided that conjunctival lesion measures ≥1 cm in diameter by tape measure and is documented by photo or there are multiple conjunctival lesions measuring together >1.5 cm. At least one of the lesions needs be histologically confirmed as EMZL.
7. Participants must be willing to provide tissue biopsy from the most recent available archival tissue or undergo an incisional or excisional lymph node or tissue biopsy. If biopsy can be reviewed to confirm the diagnosis but there is no extra tissue for exploratory studies, such participants can still be enrolled in this trial.
8. Participant should have at least one of the following criteria for treatment initiation:

   * Threatened extranodal organ function
   * Involvement of ≥3 nodal sites, each with diameter of ≥3 cm
   * Any nodal or extranodal tumor mass with a diameter of ≥5 cm
   * B symptoms (fever ≥38 degrees Celsius of unclear etiology, night sweats, weight loss >10% within the prior 6 months) or other symptoms attributed to disease or specific organ involvement associated with the relapse.
   * Risk of local compressive symptoms that may result in organ compromise
   * Splenomegaly or splenic lesion without splenomegaly
   * Leukopenia attributed to MZL (leukocytes <1000/mm3)
   * Leukemia (>5,000 lymphoma cells/mm3)
   * Requirement for transfusion or growth factor support attributed to lymphoma
   * Involvement of 2 or more extranodal sites, with tumor/lesion in each extranodal site ≥1 cm
9. Life expectancy >3 months.
10. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
11. Adequate hematologic, hepatic, and renal function tested within 6 weeks prior to the start of therapy (values must not be achieved with growth factors):

    * Absolute neutrophil count (ANC) ≥1.0 × 10^9/L.
    * Hemoglobin ≥8.0 g/dL.
    * Platelet count ≥ 75 × 10^9/L.
    * Total bilirubin ≤1.5 × upper limit normal (ULN). Participants with documented history of Gilbert's syndrome and in whom total bilirubin elevations are accompanied by elevated indirect bilirubin are eligible.
    * Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≤3.0 × ULN or ≤5 × ULN in the presence of liver involvement by lymphoma.
    * Creatinine within normal institutional limits, or

      * calculated creatinine clearance ≥30 mL/min/1.73 m2 using the Modification of Diet in Renal Disease formula
      * calculated creatinine clearance ≥35 mL/min by the Cockcroft-Gault Equation (Cockcroft, 1976)
      * estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 using the Modification of Diet in Renal Disease formula for participants with creatinine levels above institutional normal (unless due to lymphoma)
12. Willingness to avoid pregnancy during the trial and for at least 90 days after the last dose of the trial intervention.

Exclusion Criteria:

1. Evidence of diffuse large B cell lymphoma (DLBCL) transformation. Participants with presumptive evidence of transformation based on clinical assessment of factors such as, but not limited to, increasing lactate dehydrogenase, rapidly worsening disease, or frequent B-symptoms, must be ruled out for a transformation to a more aggressive disease, such as DLBCL.
2. History of central nervous system lymphoma (either primary or metastatic) or leptomeningeal disease. Participants with Dural MZL are eligible.
3. Patients that need immediate cytoreduction.
4. Concurrent or previous anticancer therapy (eg, chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, investigational therapy, or tumor embolization).
5. Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone (>20 mg), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1.

   1. Steroids that are used for treatment of allergy or other underlying condition are permittable, but not steroids started to treat lymphoma. Participants receiving corticosteroids must be at a dose level ≤20 mg/day within 7 days of the trial intervention administration.
   2. The use of inhaled corticosteroids is permitted
   3. The use of mineralocorticoids for management of orthostatic hypotension is permitted
   4. Single dose of dexamethasone for nausea or B symptoms is permitted
   5. Antibiotic treatment of H. pylori-positive gastric EMZL is permitted
6. Allogeneic stem cell transplant, or autologous stem cell transplant or Chimeric antigen receptor T-cell therapy for any indication
7. Active graft versus host disease.
8. Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
9. Current or previous other malignancy within 3 years of trial entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.
10. Significant concurrent, uncontrolled medical condition, including, but not limited to, renal, hepatic, hematological, gastrointestinal (GI), endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
11. Chronic or current active infectious disease (including severe acute respiratory syndrome (SARS) coronavirus 2 (CoV-2)) requiring systemic antibiotics, antifungal, or antiviral treatment or any major episode of infection requiring treatment with IV antibiotics within 4 weeks of Day 1 of Cycle 1
12. Exposure to a live vaccine within 30 days of administration or anticipation that a live attenuated vaccine will be required during the study.

    1. Inactivated influenza vaccinations may be given during the influenza season.
    2. An approved coronavirus disease 2019 (COVID-19) vaccine (messenger ribonucleic acid (mRNA), inactivated virus, and replication deficient viral vector vaccines) is allowed.
13. Known human immunodeficiency virus (HIV) infection or positivity on immunoassay. Note: HIV screening test is optional
14. History of solid organ transplantation
15. History of severe allergic or anaphylactic reaction to humanized, chimeric or murine monoclonal antibodies (MAbs)
16. Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary (CHO) cells or any component of the mosunetuzumab, lenalidomide, or thalidomide formulation, including mannitol.
17. Significant cardiovascular disease (eg, New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 3 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
18. Known or suspected chronic active Epstein-Barr virus (EBV) infection
19. Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
20. History of progressive multifocal leukoencephalopathy (PML)
21. Active hepatitis B infection

    a. Patients who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive, must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation
22. Active hepatitis C infection

    a. Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation
23. History of autoimmune disease, including, but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

    1. Patients with a remote history of, or well-controlled, autoimmune disease with a treatment free interval from immunosuppressive therapy for 12 months may be eligible to enroll if judged to be safe by the investigator
    2. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible
    3. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
    4. Patients with a history of disease-related immune thrombocytopenic purpura, or autoimmune hemolytic anemia may be eligible
    5. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (eg, patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

       * i. Rash must cover 10% of body surface area
       * ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids
       * iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency oral corticosteroids within the previous 12 months
24. Positive SARS-CoV-2 test within 7 days prior to enrollment. Rapid antigen test result is also acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | Up to 12 months
  The number of participants with best overall response of complete response (CR) to protocol therapy will be reported. Response will be assessed using Cheson 2014 criteria if disease is not FDG-avid in initial screening, and by revised Lugano 2014 criteria if screening Fluorodeoxyglucose (FDG) positron emission tomography (PET) computed tomography (CT) (FDG PET/CT) demonstrated FDG-avid disease.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 months
  The number of participants with best overall response of complete response (CR) or partial response (PR) to protocol therapy will be reported. Response will be assessed using Cheson 2014 criteria if disease is not FDG-avid in initial screening, and by revised Lugano 2014 criteria if screening FDG-PET/CT demonstrated FDG-avid disease.
Partial Response (PR) Rate | Up to 12 months
  The number of participants with partial response (PR) to protocol therapy will be reported. Response will be assessed using Cheson 2014 criteria if disease is not FDG-avid in initial screening, and by revised Lugano 2014 criteria if screening FDG-PET/CT demonstrated FDG-avid disease.
Number of Participants Experiencing treatment-related adverse events | Up to 13 months
  The number of participants experiencing toxicity will be reported as the number of participants experiencing treatment-related adverse events (AEs), and serious adverse events (SAEs) regardless of attribution. Toxicity will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Number of Participants Experiencing Cytokine Release Syndrome Adverse Events | Up to 13 months
  The number of participants experiencing cytokine release syndrome (CRS) related adverse events (AEs) will be reported. CRS AEs will be assessed according to the American Society for Transplantation and Cellular Therapy (ASTCT) Consensus 2019 Grading Criteria.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is the elapsed time from start of treatment to documented progressive disease or death from any cause. For participants alive and progression-free, follow-up will be censored at the last date of document progression-free status.
Time to Response (TTR) | Up to 2 years
  Time to response (TTR) is defined as elapsed time from start of treatment to achievement of complete response (CR) or partial response (CR).
Duration of Response (DOR) | Up to 2 years
  Duration of response (DOR) is the elapsed time from achievement of objective response (CR or PR) to progression, relapse, or death from any cause.
Overall Survival (OS) | Up to 3 years
  Overall survival (OS) is the elapsed time from start of treatment to death from any cause. Alive participants will be censored at last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Izidore Lossos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No